CLINICAL TRIAL: NCT04720339
Title: Molecular Monitoring of cfDNA by ddPCR in Non-small Cell Lung Cancer Treated by Immunotherapy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7652
Record Dates: First submitted 2020-02-12; First posted 2021-01-22 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: NSCLC; IMMUNOTHERAPY; QUANTIFICATION OF CELL-FREE DNA
Keywords: NSCLC; Cell-free DNA; Immunotherapy; Digital PCR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Genetic: Molecular monitoring by quantification of cell-free DNA

INTERVENTIONS:
Genetic: Molecular monitoring by quantification of cell-free DNA — Molecular monitoring by quantification of cell-free DNA (absolute value and variation from baseline) of two house-keeping genes (RPP30, TMEM11) by droplet digital PCR, during based-immunotherapy treatments of NSCLC patients.
  Cell-free DNA will be extracted from 4 ml of plasma before treatments by immunotherapy, obtained from blood Streck® tubes.
  Quantification of house-keeping genes (or mutated genes if some are previously routinely identified in tumor tissue) by ddPCR.

SUMMARY:
Non-small cell lung cancer (NSCLC) is a major public health problem. New treatments as immunotherapy can improve prognosis of patients with NCLC tumors. Nevertheless, no robust biomarker is actually available.

The hypothesis of the trial is to realize a longitudinal molecular monitoring of NSCLC patients treated by immunotherapy using a quantitative analysis of cell-free DNA.

The primary purposes is to study the predictive value of quantification of cell-free DNA at the first reevaluation time, on the clinical benefit, in NSCLC patients treated by immunotherapy (regardless of line, or associated treatments) The secondary purposes in this population of patients is to study the earlier predictive value (before the second treatment by immunotherapy ) of quantification of cell-free DNA, and its relationship with refractory disease and pseudo-progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* informed of the objectives of the project and signed consent
* non small cell lung cancer, stage IIIA, IIIB or IV
* PS (WHO performance status) < or =2
* treatment based on immunotherapy (monotherapy or combination)
* at least one measurable target
* available results of PD-L1 expression

Exclusion Criteria:

* concomitant other type of cancer
* another cancer in the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2025-05-27 (Estimated); Study Completion 2027-10-27 (Estimated)

PRIMARY OUTCOMES:
Predictive value of quantification of cell-free DNA from plasma at the time of the first radiological evaluation, on clinical benefit | Inclusion visit - visit 2 (day 60)
  The quantification of cell-free DNA is realized by droplet digital PCR (ddPCR) using two house-keeping genes (RPP30, TMEM11); if a somatic mutation is identified in the paired tumor DNA in routine practice, this mutation is also quantify in the cell-free DNA from plasma. The quantification of cell-free DNA corresponds to the variation from the time at inclusion and the time at the first radiological evaluation.
  The clinical benefit is defined by the duration of treatment by immunotherapy.

SECONDARY OUTCOMES:
Study of the earlier predictive value (before the second treatment by immunotherapy ) of quantification of cell-free DNA, and its relationship with refractory disease and pseudo-progressive disease. | Inclusion visit, visit 1 (day 15), visit 2 (day 60), visit 3 (day 180), visit 4 (day 270), visit 5 (day 360), visit 6 (day 720), or early termination visit (in case of progression with end of immunotherapy)
  The quantification of cell-free DNA is realized by droplet digital PCR (ddPCR) using two house-keeping genes (RPP30, TMEM11); if a somatic mutation is identified in the paired tumor DNA in routine practice, this mutation is also quantify in the cell-free DNA from plasma.
  The earlier quantification of cell-free DNA corresponds to the variation from the time at inclusion and the time before the second administration of immunotherapy.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU de Besancon - Service de pneumologie, Besançon
  - Hopitaux Civils de Colmar - service de Pneumologie, Colmar
  - CHU de Dijon - service de Pneumologie, Dijon
  - CLCC Georges-François Leclerc, Dijon
  - GHR Mulhouse Sud-Alsace - Service de Pneumologie, Mulhouse
  - CHU de Reims - service de Pneumologie, Reims
  - CHRU de Strasbourg, Strasbourg
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No